CLINICAL TRIAL: NCT00002478
Title: Phase II Study of Prolonged Oral VP-16 for Advanced Ovarian Epithelial and Cervical Cancer
Brief Title: Etoposide in Treating Patients With Advanced Ovarian or Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000077078; GOG-26LL
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2000-11

CONDITIONS: Cervical Cancer; Ovarian Cancer
Keywords: recurrent cervical cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Etoposide

INTERVENTIONS:
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of etoposide in treating patients who have refractory, recurrent, or metastatic ovarian or cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of prolonged oral etoposide (VP-16) in patients with advanced ovarian epithelial or cervical cancer. II. Evaluate the frequency and severity of observed adverse effects in this patient population treated with prolonged oral VP-16.

OUTLINE: Patients receive etoposide by mouth once daily on days 1-21 every 4 weeks. Patients with responding disease continue treatment for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients with stable disease continue treatment for up to 6 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: If 4-6 responses are observed in the first 25 patients, an additional 15 patients will be entered. The estimated duration of the study is 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or metastatic ovarian epithelial or cervical cancer Tissue not accessible for biopsy Refractory to curative therapy or established treatments and ineligible for higher priority GOG protocols Measurable disease required, as follows: Lesion measurable by physical exam Lesion bidimensionally measurable on sonogram or imaging Ascites/pleural effusion not measurable

PATIENT CHARACTERISTICS: Age: Any age Performance status: GOG 0-2 Hematopoietic: WBC at least 3,000/mm3 Absolute granulocyte count at least 1,500/mm3 Platelets at least 100,000/mm3 Hepatic: Bilirubin no more than 1.5 times normal AST no more than 3 times normal Alkaline phosphatase no more than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Other: Body surface area at least 1 square meter No requirement for intravenous hydration or nutritional support No significant infection No second malignancy other than nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since anticancer therapy Chemotherapy: No more than 1 prior chemotherapy trial No prior etoposide At least 3 weeks since chemotherapy and recovered Endocrine therapy: At least 3 weeks since anticancer therapy Radiotherapy: At least 3 weeks since radiotherapy Surgery: At least 3 weeks since surgery and recovered

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-06; Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Study Chair — University Hospitals Seidman Cancer Center
Locations (47):
- United States (47):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Result] Rose PG, Blessing JA, Buller RE, Mannel RS, Webster KD. Prolonged oral etoposide in recurrent or advanced non-squamous cell carcinoma of the cervix: a Gynecologic Oncology Group study. Gynecol Oncol. 2003 May;89(2):267-70. doi: 10.1016/s0090-8258(03)00079-9. PMID 12713990
- [Result] Rose PG, Blessing JA, Mayer AR, Homesley HD. Prolonged oral etoposide as second-line therapy for platinum-resistant and platinum-sensitive ovarian carcinoma: a Gynecologic Oncology Group study. J Clin Oncol. 1998 Feb;16(2):405-10. doi: 10.1200/JCO.1998.16.2.405. PMID 9469322
- [Result] Kudelka A, ed.: A phase II study of prolonged oral VP-16 in women with refractoy epithelial ovarian carcinoma. [Abstract] Proceedings of the American Society of Clinical Oncology 13: A-888, 276, 1994.